CLINICAL TRIAL: NCT00171418
Title: Assessment of the Effects of Tegaserod in the Management of Gastroesophageal Reflux Disease (GERD) in Patients With Incomplete Response to Proton Pump Inhibitors (PPIs).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHTF919BUS26
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; PPI
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Study to assess the effects of adding tegaserod to PPI therapy results in clinically meaningful improvement of GERD symptoms in patients with incomplete relief of symptoms on daily PPI therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* GERD symptoms for at least 6 months
* PPI therapy for at least 4 weeks
* Incomplete symptom relief on daily PPI therapy
* No erosive disease as evidenced in EGD/no change in symptom severity

Exclusion Criteria:

* Evidence of structural abnormality of the gastrointestinal tract or disease/conditions
* Previous gastrointestinal surgery that may influence esophageal motor function
* Known primary esophageal motor disorder other than Inefficient Esophageal Motor Disorder
* Evidence of cathartic colon or a history of laxative use

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2003-06; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To determine the effect of 4 weeks of tegaserod treatment in addition to PPI on clinically meaningful incremental gain in improvement of overall GERD symptoms, based on weekly binary questions.

SECONDARY OUTCOMES:
To evaluate the sensitivity of three global symptom assessments, including two binary scales and a Likert-type scale along with a composite symptom index (end of treatment compared to baseline)
To evaluate frequency, severity and bothersomeness of individual GERD symptoms (daily assessments)
Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (2):
- United States (2):
  - Drug Research Services, Inc, Metairie, Louisiana
  - The Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma